CLINICAL TRIAL: NCT00505791
Title: Double Blind Randomized Placebo Controlled Trial of Natrecor in Patients Hospitalized for Decompensated Heart Failure in the Presence of a Normal Left Ventricular Ejection Fraction
Brief Title: Double Blind Randomized Placebo Controlled Trial of Natrecor in Acute Decompensated Heart Failure With Normal EF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll patients
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0120050150; IRB # 0120050150 (Other Grant/Funding Number: UMDNJ 106199)
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure, Congestive; Dyspnea; Pulmonary Edema
Keywords: Acute decompensated heart failure; Normal left ventricular ejection fraction; Vasodilator therapy
MeSH Terms: conditions — Heart Failure; Dyspnea; Pulmonary Edema | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator): Lactose, NF (monohydrate)
  Interventions: Drug: Nesiritide
- Nesiritide (Active Comparator): Natrecor (nesiritide) is a commercially available B-type natriuretic peptide which is indicated for intravenous treatment of patients with acutely decompensated congestive heart failure who have dyspnea at rest or with minimal activity.
  Interventions: Drug: Nesiritide

INTERVENTIONS:
Drug: Nesiritide — Study drug will be administered for 24 hours. Study drug will be initiated with a 2-µg/kg loading bolus followed by .01-µg/kg/min infusion. This may be increased at a rate of .005-µg/kg/min. every 3 hours until maximum dose of .03-µg/kg/min. Any increase in the infusion rate will be preceded by a 1-µg/kg bolus and increases in infusion rates will be permitted only in patients who have a systolic blood pressure > 100 mmHg.
  Other Names: Natrecor

SUMMARY:
Heart failure (HF) is a disease that is caused by a reduced heart muscle function. Reduced heart muscle function can occur as a consequence of reduced pumping activity from a weak heart muscle or because of a stiff heart muscle. This study is looking at the effectiveness of Natrecor (nesiritide) in patients that require hospitalization due to worsening heart failure as a result of a stiff or thickened heart muscle. Natrecor is a man-made version of a protein that my body makes on its own and has been approved for the treatment of patients requiring hospital admission for heart failure and have shortness of breath at rest or with minimal activity.

Natrecor has shown to lower the pressures in the heart and decreases the congestion in the lungs. This study is being done to see if the addition of a Natrecor to standard medical therapy for HF will improve symptoms faster or more completely than giving only the standard treatment for CHF.

DETAILED DESCRIPTION:
Despite an increasing number of patients hospitalized with decompensated heart failure in the presence of a normal ejection fraction, there is little clinical trial data to guide clinicians in their acute management . Since the number of patients hospitalized with decompensated heart failure in the presence of normal ejection fraction (>50%) is increasing, it is imperative to develop effective therapies which are supported by clinical evidence such as randomized clinical trials. The purpose of this study is to evaluate the utility of natriuretic peptide for the specific management of these patients.

Loop diuretics (such as Furosemide) are powerful diuretic agents which are used as a first-line therapy in volume overloaded patients with low ejection fraction heart failure. Despite their widespread use, they can cause severe electrolyte and volume abnormalities contributing to increased morbidity and mortality . These adverse effects are exacerbated even further in heart failure patients with normal ejection fraction since these patients are usually older, have worse renal function and are more susceptible to volume depletion and its effects. The FDA approved Natrecor for Acute Decompensated Heart Failure and did not differ between low ejection fraction and normal ejection fraction heart failure. Given however, the low number of patients with normal ejection fraction heart failure in clinical trials and the paucity of outcome data in these patients, we propose to specifically study them.

Brief Description of Experimental Approach:

Patients who present to the emergency room diagnosed with acute decompensated heart failure requiring the administration of intravenous diuretics and found to have normal contractile function will be eligible for participation in this study. Patients must have pulmonary congestion documented on their admitting chest X-ray and clinical evidence of volume overload such as rales or edema on physical examination at the time of randomization. Patients will have received at least one dose of IV Furosemide either in-route to the emergency room or on presentation to the emergency room. An echocardiogram will be obtained after presentation to the emergency room documenting a normal (>50%) left ventricular ejection fraction. Patients will be randomized to Natrecor or placebo in addition to a standard medical therapy. Study drug will be administered for 24 hours. Study drug will be initiated with a 2-µg/kg loading bolus followed by .01-µg/kg/min infusion. This may be increased at a rate of .005-µg/kg/min. every 3 hours until maximum dose of .03-µg/kg/min. Any increase in the infusion rate will be preceded by a 1-µg/kg bolus and increases in infusion rates will be permitted only in patients who have a systolic blood pressure > 100 mmHg. IV Nitroglycerin and IV Milrinone will be prohibited within 2 hours prior to initiating study drug infusion to three hours after completion of study drug infusion. All other intravenous vasoactive medications including other IV inotropes will be avoided within 2 hours prior to initiating study drug infusion to three hours after start of study drug infusion. Oral ACE inhibitors will be avoided from 2 hours prior to initiating study drug infusion to 30 minutes after start of study drug so as to avoid potential hypotension. Concomitant 'standard of care medications' including diuretics (IV or PO), ACE inhibitors, Aldactone, Digoxin etc. will be left to investigator discretion to be administered during the hospital stay as indicated. The primary endpoint of this study will be an absolute reduction in brain natriuretic peptide (BNP) levels three hours after discontinuation of the study drug. BNP is elevated in acute decompensated heart failure and has utility in outcome, severity and prognosis of patients with ADHF .

Secondary endpoints will include: all cause in-hospital mortality, physician and patient global score at 24 hours, twenty-four hour urine output after start of study drug infusion, weight change at 24 hours after start of study drug infusion, number of patients with K < 3.5meq at 24 hours, change in creatinine at 24 hours after start of study drug and at discharge or at 3 days, BNP levels at baseline, 3 hours after discontinuation of the study drug and at discharge or at 3 days, total diuretic dose of IV and PO Lasix at 48 hours and 72 hours after randomization or at discharge, changes in diastolic indices measured by transthoracic echocardiography 24 hours after the start of the study drug and 30 day post-randomization all cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years of age
* Admission to the ED for congestive heart failure requiring IV diuretics and hospitalization
* Chest X-ray evidence of pulmonary congestion (pleural effusion will not suffice).
* Physical evidence of volume overload i.e. rales or edema at time of randomization.
* Normal left ventricular ejection fraction (EF >50%) on echocardiography after presentation to the ER.
* Patients must be able to provide informed consent.

Exclusion Criteria:

* Acute coronary syndrome with evidence of active ischemia as evident by acute ST segment or T wave changes or initial cardiac enzymes that demonstrate myocardial necrosis or requiring IV nitroglycerin for treatment.
* Hemodynamically unstable patients that require invasive monitoring or mechanical ventilation.
* Cardiogenic shock, volume depletion, or any other clinical condition that would contraindicate the administration of IV diuretics, ACE inhibitors, or an IV agent with potent vasodilating properties.
* Systolic blood pressure >220mmHg or diastolic blood pressure >110mHg.
* Systolic blood pressure consistently <90 mmHg.
* Tachyarrhythmia (HR>120).
* Bradyarrythmia (HR < 50).
* Myocarditis.
* Hypertrophic obstructive cardiomyopathy.
* Restrictive or infiltrative cardiomyopathy including amyloid or sarcoid.
* Constrictive cardiomyopathy.
* Primary right sided heart failure or severe pulmonary hypertension (pulmonary artery pressure > 60mmHg).
* Significant aortic or mitral valve stenosis (Aortic Valve Area < 1.0cm2, Mitral Valve Area < 1.5 cm2 ).
* Aortic or mitral insufficiency ≥ 3+.
* Malfunctioning artificial valve.
* Uncorrected congenital heart disease.
* Concomitant administration of IV Dobutamine, or other IV vasoactive medications from 2 hours before the start of the study drug until 3 hours after the start of the study drug;
* Administration of IV Nitroglycerin or IV Milrinone.
* Concomitant administration of oral ACE inhibitor medication from 2 hours before the start of the study drug until 30 minutes after the start of the study drug.
* Severe COPD/Asthma as assessed by clinical criteria, prior PFT's or if the patient requires chronic oral steroid treatment.
* Other significant pulmonary disease that causes significant SOB/DOE i.e. pneumoconiosis etc.
* Patients with creatinine > 3.0 mg/dl.
* Patients with a serum potassium level < 3.5, >5.5 mmol/l.
* Anemia with a Hob < 9 g/dl.
* Acute neurological event.
* Known allergic reaction or contraindication to Natrecor or furosemide.
* Pregnancy or suspected pregnancy.
* Patients with a history of ETOH abuse or other illicit drug abuse.
* Patients with active liver, hematologic, gastrointestinal, immunologic, endocrine, metabolic, central nervous system or other medical condition disease which in the opinion of the investigator may adversely effect the safety and efficacy of the study drug or the lifespan of the patient.
* Therapy with an investigational drug.
* Unwillingness or inability to comply with study requirements including the 30-day follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study will be an absolute reduction in brain natriuretic peptide (BNP) three hours after discontinuation of the study drug. | Three hours after discontinuation of the study drug

SECONDARY OUTCOMES:
All cause in-hospital mortality | 30 days post-randomization
Physician and patient global score at 24 hours | 30 days post-randomization
Twenty-four hour urine output after start of study drug infusion | 30 days post-randomization
Weight change at 24 hours after start of study drug infusion | 30 days post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Marc Klapholz, MD, Principal Investigator — University of Medicine and Dentistry of New Jersey/ New Jersey Medical School
Locations (1):
- University of Medicine and Dentistry of New Jersey/ New Jersey Medical School, Newark, New Jersey, United States

REFERENCES:
- [Background] Polanczyk CA, Rohde LE, Dec GW, DiSalvo T. Ten-year trends in hospital care for congestive heart failure: improved outcomes and increased use of resources. Arch Intern Med. 2000 Feb 14;160(3):325-32. doi: 10.1001/archinte.160.3.325. PMID 10668834
- [Background] Publication Committee for the VMAC Investigators (Vasodilatation in the Management of Acute CHF). Intravenous nesiritide vs nitroglycerin for treatment of decompensated congestive heart failure: a randomized controlled trial. JAMA. 2002 Mar 27;287(12):1531-40. doi: 10.1001/jama.287.12.1531. PMID 11911755
- [Background] Francis GS, Siegel RM, Goldsmith SR, Olivari MT, Levine TB, Cohn JN. Acute vasoconstrictor response to intravenous furosemide in patients with chronic congestive heart failure. Activation of the neurohumoral axis. Ann Intern Med. 1985 Jul;103(1):1-6. doi: 10.7326/0003-4819-103-1-1. PMID 2860833
- [Background] Weinfeld MS, Chertow GM, Stevenson LW. Aggravated renal dysfunction during intensive therapy for advanced chronic heart failure. Am Heart J. 1999 Aug;138(2 Pt 1):285-90. doi: 10.1016/s0002-8703(99)70113-4. PMID 10426840
- [Background] Mueller C, Scholer A, Laule-Kilian K, Martina B, Schindler C, Buser P, Pfisterer M, Perruchoud AP. Use of B-type natriuretic peptide in the evaluation and management of acute dyspnea. N Engl J Med. 2004 Feb 12;350(7):647-54. doi: 10.1056/NEJMoa031681. PMID 14960741
- [Background] Butler J, Emerman C, Peacock WF, Mathur VS, Young JB; VMAC study investigators. The efficacy and safety of B-type natriuretic peptide (nesiritide) in patients with renal insufficiency and acutely decompensated congestive heart failure. Nephrol Dial Transplant. 2004 Feb;19(2):391-9. doi: 10.1093/ndt/gfg558. PMID 14736964